CLINICAL TRIAL: NCT00635466
Title: Phase II Trial to Evaluate Laparoscopic Surgery for Stage 0/I Rectal Carcinoma
Acronym: Lap RC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Japan Society of Laparoscopic Colorectal Surgery (Network)
Responsible Party: Masahiko Watanabe, Kitasato University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lap RC; NCCHCT19-49
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Rectal Cancer
Keywords: laparoscopic surgery, rectal carcinoma, phase II trial
MeSH Terms: conditions — Rectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lap, 1 (Experimental): Patients undergoing laparoscopic surgery for rectal carcinoma
  Interventions: Procedure: laparoscopic surgery for rectal carcinoma

INTERVENTIONS:
Procedure: laparoscopic surgery for rectal carcinoma — Laparoscopic resection of the rectum with adequate lymphadenectomy is performed according to the General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus edited by the Japanese Society for Cancer of the Colon and Rectum. The extent of lymphadenectomy and site of ligation and division of the inferior mesenteric vessels were decided by the surgeon in charge. Pneumoperitoneal approaches are used to explore the abdomen, mobilize the left side colon, identify critical structures and ligate the vascular pedicle. Mobilization of the rectum, excision of the mesorectum, rectal transection, removal of the specimen, and reconstruction are performed by the pneumoperitoneal approach or the extracorporeal approach via a small incision (<8 cm).
  Other Names: laparoscopic rectal resection

SUMMARY:
The purpose of this study is to examine the technical and oncological feasibility of laparoscopic surgery for rectal carcinoma

DETAILED DESCRIPTION:
Recently reported randomized controlled trials demonstrated that laparoscopic surgery was comparable or superior to open surgery regarding the long-term outcome for colon and rectosigmoidal carcinoma; however, controversy persists regarding the appropriateness of laparoscopic surgery for patients with rectal carcinoma because of the uncertainty of the long-term outcome, and of concerns over the safety of the procedure. In Japan, lateral lymph node dissection combined with total mesorectal excision remains the standard surgical procedure for patients with advanced lower rectal carcinoma, and lateral lymph node dissection by laparoscopy is still an unexplored frontier. To examine the technical and oncological feasibility of laparoscopic surgery for rectal carcinoma, a phase II trial will be conducted in patients with a preoperative diagnosis of stage 0/I rectal carcinoma, under the direction of the Japan Society of Laparoscopic Colorectal Surgery, to which leading hospitals in laparoscopic surgery for colorectal carcinoma in Japan are members.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven rectal carcinoma.
2. Tumor located in the rectum.
3. Clinical Tis, T1, T2 N0 M0
4. Without multiple lesions other than carcinoma in situ
5. Tumor size <8 cm.
6. Sufficient organ function.
7. No bowel obstruction.
8. No history of major colorectal surgery.
9. No history of chemotherapy or radiotherapy.
10. Provide written informed consent.

Exclusion Criteria:

1. Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ.
2. Pregnant or lactating women.
3. Severe mental disease.
4. Severe pulmonary emphysema, interstitial pneumonitis or ischemic heart disease.
5. Continuous systemic steroid therapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2008-02; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year

SECONDARY OUTCOMES:
anastomotic leakage rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Masahiko Watanabe, PhD, Study Chair — Kitasato University Hospital
Locations (1):
- Kitasato University Hospital, Sagamihara, Kanagawa, Japan

REFERENCES:
- [Background] Yamamoto S, Yoshimura K, Konishi F, Watanabe M. Phase II trial to evaluate laparoscopic surgery for Stage 0/I rectal carcinoma. Jpn J Clin Oncol. 2008 Jul;38(7):497-500. doi: 10.1093/jjco/hyn054. Epub 2008 Jun 26. PMID 18586667
- [Derived] Ito M, Yamamoto S, Okuda J, Fujii S, Yamaguchi S, Otsuka K, Yoshimura K, Watanabe M; Japan Society of Laparoscopic Colorectal Surgery. Long-term survival outcomes following laparoscopic surgery for clinical stage 0/I rectal carcinoma. Ann Gastroenterol Surg. 2020 May 20;4(3):294-300. doi: 10.1002/ags3.12333. eCollection 2020 May. PMID 32490343
- [Derived] Yamamoto S, Ito M, Okuda J, Fujii S, Yamaguchi S, Yoshimura K, Sugihara K, Watanabe M; Japan Society of Laparoscopic Colorectal Surgery. Laparoscopic surgery for stage 0/I rectal carcinoma: short-term outcomes of a single-arm phase II trial. Ann Surg. 2013 Aug;258(2):283-8. doi: 10.1097/SLA.0b013e318283669c. PMID 23426337
- See also: Click here for the information regarding the Japanese Society for Cancer of the Colon and Rectum (JSCCR). — http://www.jsccr.jp/